CLINICAL TRIAL: NCT01038557
Title: Efficacy and Safety of Frozen Red Blood Cells for Transfusion in Trauma Patients
Brief Title: Frozen Red Blood Cell Transfusions in Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: United States Air Force (U.S. Federal Agency); Armed Services Blood Program (Unknown)
Responsible Party: Principal Investigator, Martin A Schreiber, MD, Professor & Chief of Trauma, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002-01
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Blood Loss; Anemia; Trauma
Keywords: frozen; red blood cells; transfusion; trauma
MeSH Terms: conditions — Hemorrhage; Anemia; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Refrigerated RBCs 0-14 days old (Active Comparator): Standard, refrigerated RBC units stored up to 14 days
  Interventions: Biological: RBC units
- Refrigerated RBCs 15-42 days old (Active Comparator): Standard, refrigerated RBC units stored 15-42 days
  Interventions: Biological: RBC units
- Frozen RBCs (Experimental): RBC units stored frozen at -80 degrees Celsius, then thawed and deglycerolized using the ACP 215.
  Interventions: Biological: RBC units

INTERVENTIONS:
Biological: RBC units — When a transfusion is ordered, enrolled subjects will receive RBC units 1) up to 14 days old, 2) 14-42 days old, or 3) that are frozen when stored.

SUMMARY:
The purpose of this study is to look at red blood cell (RBC) transfusions in trauma patients and evaluate for any differences between the age of the RBCs and how they were stored. The investigators will specifically look for the following differences between study groups:

1. the transfused red blood cells' ability to delivery oxygen to the tissues
2. differences in biochemical markers in subjects and units transfused, and
3. how the subject's internal organs are working and if they develop any infections

ELIGIBILITY:
Inclusion Criteria:

* Trauma Service with an Injury Severity Score > 4
* Require a blood (PRBC) transfusion
* Transfusion is not emergent
* Able to obtain consent from patient or appropriate 3rd party prior to 1st transfusion

Exclusion Criteria:

* Inability to adhere to blood age randomization due to limitations of the blood bank inventory
* Bilateral hand injuries that prevent StO2 measurements
* Age < 15
* Pregnancy
* Massive transfusion (=/> 10 units in 24 hours) in last 3 months
* Hemodynamically unstable or need for transfusion in < 3 hours

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2010-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schreiber, MD, Principal Investigator — Oregon Health and Science University
Locations (5):
- United States (5):
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Started | 82 | 86 | 86
Completed | 82 | 86 | 86
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs | Total
Number analyzed (Participants) | 82 | 86 | 86 | 254
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52.3 [29.4 to 62.5] | 47.9 [28.1 to 67.0] | 49.3 [30.9 to 62.6] | 49.3 [29.4 to 62.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 40 | 29 | 101
  Male | 50 | 46 | 57 | 153
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 82 | 86 | 86 | 254
Injury Severity Score [Median (Inter-Quartile Range); unit: units on a scale (1 best to 75 worst)] | 19 [10 to 32] | 19 [11 to 26] | 19 [14 to 26] | 19 [10 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Tissue Oxygenation
Description: Assessment of tissue oxygenation by NIRS in subjects up to 3 hours after PRBC transfusion.
Time Frame: Percentage of baseline (3 hours post transfusion compared to baseline)
Population: Mean percent change in tissue oxygenation (StO2) over time is reported for subjects with continuous data. Data on subjects whose NIRS device fell off or there was discontinuity in recording were excluded.
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 76 | 73 | 82
percentage of baseline | 100.3 (7.2) | 98.2 (11.4) | 98.3 (14.1)

2. Secondary Outcome: 2,3 DPG Levels After Transfusion
Description: 2,3 DPG levels 12 hours after transfusion
Time Frame: 12 hours post transfusion
Population: Blood samples to measure 2,3 DPG levels could not be collected from all subjects 12 hours after transfusion or results were not measurable.
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 60 | 75 | 70
g/L | 0.33 [0.22 to 0.47] | 0.36 [0.25 to 0.47] | 0.31 [0.23 to 0.56]

3. Secondary Outcome: Free Hemoglobin Levels After Transfusion
Description: Free hemoglobin levels 12 hours after transfusion
Time Frame: 12 hours after transfusion
Population: Blood samples to measure free hemoglobin could not be collected from all subjects 12 hours after transfusion or the results were not measurable.
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 63 | 75 | 69
ug/mL | 201 [86 to 422] | 194 [106 to 194] | 174 [82 to 287]

4. Secondary Outcome: Haptoglobin Levels 12 Hours After Transfusion
Description: Haptoglobin levels after transfusion
Time Frame: 12 hours after transfusion
Population: Blood samples to measure haptoglobin could not be collected from all subjects 12 hours after transfusion or the results were not measurable.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 62 | 75 | 69
ng/mL | 897 [349 to 1775] | 1470 [494 to 2360] | 1350 [411 to 2700]

5. Secondary Outcome: Clinical Outcomes - Hospital Days
Description: Clinical outcomes - Number of days admitted to the hospital within a 6 month window.
Time Frame: from time of randomization through hospital discharged, assessed up to 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 82 | 86 | 86
days | 13 [8 to 20.5] | 13.5 [9 to 22] | 18 [10 to 26]

6. Secondary Outcome: Clinical Outcomes - ICU Days
Description: Number of days admitted to the ICU during hospital admission
Time Frame: from time of randomization through hospital discharged, assessed up to 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 82 | 86 | 86
days | 6 [2 to 11] | 5 [2 to 11] | 7 [3 to 14.5]

7. Secondary Outcome: Clinical Outcomes - Ventilator Days
Time Frame: from time of randomization through hospital discharged, assessed up to 6 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 82 | 86 | 86
days | 0 [0 to 4.5] | 0 [0 to 4.25] | 1 [0 to 9.5]

8. Secondary Outcome: Number of Participants With Acute Renal Failure
Description: Number of participants who developed acute renal failure while hospitalized.
Time Frame: from time of randomization through hospital discharged, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 82 | 85 | 86
Participants | 7 | 7 | 10

9. Secondary Outcome: Clinical Outcomes - Acute Respiratory Distress Syndrome
Description: Number of subjects who developed acute respiratory distress syndrome while hospitalized.
Time Frame: from time of randomization through hospital discharged, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 82 | 85 | 86
Participants | 5 | 2 | 4

10. Secondary Outcome: Clinical Outcomes - Infections
Description: Number of subjects who developed infections while hospitalized.
Time Frame: from time of randomization through hospital discharged, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
Number analyzed (Participants) | 82 | 85 | 86
Participants | 24 | 22 | 24

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the patient's hospital admission, up to 6 months.
Arm/Group | Refrigerated RBCs 0-14 Days Old | Refrigerated RBCs 15-42 Days Old | Frozen RBCs
All-Cause Mortality (participants affected / at risk) | 3/82 | 3/86 | 3/86
Serious Adverse Events (participants affected / at risk) | 5/82 | 6/86 | 8/86
Other Adverse Events (participants affected / at risk) | 24/82 | 22/85 | 24/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refrigerated RBCs 0-14 Days Old (N=82) | Refrigerated RBCs 15-42 Days Old (N=86) | Frozen RBCs (N=86)
Pulmonary Embolism (General disorders) | 3 (3) | 6 (6) | 5 (5) — Pulmonary Embolism
Sepsis (General disorders) | 5 (5) | 6 (6) | 8 (8) — Sepsis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Refrigerated RBCs 0-14 Days Old (N=82) | Refrigerated RBCs 15-42 Days Old (N=85) | Frozen RBCs (N=86)
Infection (Infections and infestations) | 24 (24) | 22 (22) | 24 (24) — All infections
Deep Vein Thrombosis (General disorders) | 14 (14) | 13 (13) | 14 (14) — Deep Vein Thrombosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No